CLINICAL TRIAL: NCT05032703
Title: Effect of Arm Ergometer Versus Stabilization Exercises on Trunk Control and Upper Extremity Functions in Children With Diplegia
Brief Title: Arm Ergometer Versus Stabilization Exercises on Trunk Control and Upper Extremity Functions in cp
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Reham Nafea Mohie El Din, Dr Reham Nafea master degree, faculty of physical therapy, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Arm ergometer in Cp
Record Dates: First submitted 2021-08-31; First posted 2021-09-02 (Actual); Last update posted 2023-08-31 (Actual); Status verified 2023-08

CONDITIONS: Spastic Diplegia
Keywords: Cerebral palsy / Arm ergometer
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Who Masked: Participant
Masking Description: Single blind
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm ergometer (Experimental): Children in group I will receive strength-endurance protocol of arm ergometer for 30 minutes in addition to the conventional physical therapy program for 30 minutes, per session, three times a week, for three consecutive months.
  Interventions: Device: Arm ergometer
- Trunk stabilization exercise (Experimental): Children in group II will receive trunk stabilization exercises for 30 minutes in addition to the conventional physical therapy program for 30 minutes, per session, three times a week, for three consecutive months.
  Interventions: Device: Arm ergometer

INTERVENTIONS:
Device: Arm ergometer — The conventional physical therapy program included three sets of exercises as follows:
  Flexibility exercises to restore joint mobility of soft tissues. Static and dynamic balance exercise. Functional walking exercises.
  Other Names: Stabilization exercises on BOSU ball

SUMMARY:
The purposes of the current study are to:

Define and compare between the efficacy of arm ergometer versus stabilization exercises on trunk control, hand grip power and upper limb quality of functions in children with diplegia.

DETAILED DESCRIPTION:
Studies have shown that the cycle ergometer exercise improves several parameters, such as muscle strength and endurance, along with torso control in sitting position. However, these results are presented only in a small sample. Studies with the use of cycle ergometer in the population with CP are still few and present little information about the physiological effects .Previous studies on children with CP focused on the effect of ergometer on the upper and lower extremities functions. Limited literature is available regarding the effect of arm ergometer on trunk control among this population. The current study will be carried out to define the effect of arm ergometer versus stabilization exercises on trunk control, hand grip power, upper limb function in children with diplegia.

ELIGIBILITY:
Inclusion Criteria:

1. Age ranges from six to ten years.
2. Grade of spasticity 1 to 2 according to Modified Ashworth scale.
3. Level II and III according to gross motor functional classification system.
4. Level I-III according to manual ability classification system.
5. Able to follow verbal commands and instructions included in both test and training.

Exclusion Criteria:

1. Significant visual or auditory problems according to medical reports (audio-vestibular and ophthalmic examination).
2. Structural or fixed soft tissue deformities of the upper extremities.
3. Neurological or orthopedic surgery in the past 12 months in the upper extremities.
4. Botox injection in the upper extremities in the past 6 months.

Ages: 6 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 42 (Actual)
Dates: Start 2021-11-18 (Actual); Primary Completion 2023-04-18 (Actual); Study Completion 2023-05-25 (Actual)

PRIMARY OUTCOMES:
Trunk control | 30 minutes
  Trunk control measurement scale includes 15 items that assess two main components of trunk control: static and dynamic sitting balance. While the total score is between 0 and 58, higher scores indicate a better level of performance.
Upper extremity functions | 30/45 minutes
  Quality of upper extremity scale test which consist 34 items in four main domains: dissociated movement, grasp, protective extension, and weight bearing.

SECONDARY OUTCOMES:
Hand grip strength | 5 minutes
  Hand held dynamometer used to measure muscle strength of the arm and hand in children with spastic CP. It is used to measure strength; maximal voluntary isometric contraction; objectively in kilograms, pounds or newtons.

CONTACTS AND LOCATIONS:
Overall Officials: Amira M Abd El Monem, Prof.dr, Study Chair — Cairo University; Amira F Hamed, Dr, Study Director — Cairo University; Ahmed R Abdel Fadil, Dr, Study Director — University of Alexandria
Locations (1):
- Faculty of physical therapy - Cairo university, Giza, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ashwal S, Russman BS, Blasco PA, Miller G, Sandler A, Shevell M, Stevenson R; Quality Standards Subcommittee of the American Academy of Neurology; Practice Committee of the Child Neurology Society. Practice parameter: diagnostic assessment of the child with cerebral palsy [RETIRED]: report of the Quality Standards Subcommittee of the American Academy of Neurology and the Practice Committee of the Child Neurology Society. Neurology. 2004 Mar 23;62(6):851-63. doi: 10.1212/01.wnl.0000117981.35364.1b. PMID 15037681
- [Background] Baunsgaard CB, Nissen UV, Christensen KB, Biering-Sorensen F. Modified Ashworth scale and spasm frequency score in spinal cord injury: reliability and correlation. Spinal Cord. 2016 Sep;54(9):702-8. doi: 10.1038/sc.2015.230. Epub 2016 Feb 9. PMID 26857270
- [Background] Garcia CC, Alcocer-Gamboa A, Ruiz MP, Caballero IM, Faigenbaum AD, Esteve-Lanao J, Saiz BM, Lorenzo TM, Lara SL. Metabolic, cardiorespiratory, and neuromuscular fitness performance in children with cerebral palsy: A comparison with healthy youth. J Exerc Rehabil. 2016 Apr 26;12(2):124-31. doi: 10.12965/jer.1632552.276. eCollection 2016 Apr. PMID 27162775
- [Background] Paulson A, Vargus-Adams J. Overview of Four Functional Classification Systems Commonly Used in Cerebral Palsy. Children (Basel). 2017 Apr 24;4(4):30. doi: 10.3390/children4040030. PMID 28441773
- [Background] dos Santos LJ, de Aguiar Lemos F, Bianchi T, Sachetti A, Dall' Acqua AM, da Silva Naue W, Dias AS, Vieira SR. Early rehabilitation using a passive cycle ergometer on muscle morphology in mechanically ventilated critically ill patients in the Intensive Care Unit (MoVe-ICU study): study protocol for a randomized controlled trial. Trials. 2015 Aug 28;16:383. doi: 10.1186/s13063-015-0914-8. PMID 26314881
- [Background] Scholtes VA, Becher JG, Comuth A, Dekkers H, Van Dijk L, Dallmeijer AJ. Effectiveness of functional progressive resistance exercise strength training on muscle strength and mobility in children with cerebral palsy: a randomized controlled trial. Dev Med Child Neurol. 2010 Jun;52(6):e107-13. doi: 10.1111/j.1469-8749.2009.03604.x. Epub 2010 Feb 12. PMID 20132136
- [Background] Unger M, Jelsma J, Stark C. Effect of a trunk-targeted intervention using vibration on posture and gait in children with spastic type cerebral palsy: a randomized control trial. Dev Neurorehabil. 2013;16(2):79-88. doi: 10.3109/17518423.2012.715313. PMID 23477461